CLINICAL TRIAL: NCT02281838
Title: The Intracerebral Hemorrhage Acutely Decreasing Arterial Pressure Trial II
Acronym: ICH-ADAPT II
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow enrolment after publication of the Interact III study
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Version 2.0
Record Dates: First submitted 2014-10-29; First posted 2014-11-04 (Estimated); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Intracerebral Hemorrhage
Keywords: Stroke; Hypertension
MeSH Terms: conditions — Cerebral Hemorrhage; Stroke; Hypertension | interventions — Labetalol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Target systolic BP <140mmHg (Experimental): Systolic blood pressure will be reduced to <140 mmHg within 1 hour of randomization.
  Interventions: Drug: labetalol/hydralazine/enalapril
- Target systolic BP <180mmHg (Active Comparator): Systolic blood pressure will be reduced, to <180 mmHg within 1 hour of randomization.
  Interventions: Drug: labetalol/hydralazine/enalapril

INTERVENTIONS:
Drug: labetalol/hydralazine/enalapril — Blood pressure will be treated with intravenous labetalol (10 mg starting dose)/hydralazine (5 mg starting dose)/enalapril (1.25 mg starting dose).

SUMMARY:
The vast majority of intracerebral hemorrhage (ICH) patients present with elevated blood pressure(BP). Management of BP is controversial with two competing rationales. There is some evidence that hyperacute treatment may improve outcomes by reducing the rate of hematoma expansion. Physicians have been reluctant to reduce BP early after ICH onset, fearing reduced cerebral blood flow (CBF) will increase ischemia and increase the risk of further damage. Other confounding mediators to further ischemic injury following ICH include increased platelet activity, withdrawal of antithrombotic therapy, endothelial dysfunction, inflammation and hypercoagulability.

This study is phase II of the ICH-ADAPT study. The investigators hypothesize that aggressive antihypertensive therapy will alter the natural history of heamatoma growth, improving outcomes after Intracranial Hemorrhage (ICH). The previous phase I ICH-ADAPT study has established the safety of early BP treatment.

The investigators have designed a phase II study in which ICH patients are randomized to aggressive versus conservative BP treatment using a deferred consent procedure. An adaptive randomization will be used to treat BP to < 140 mmHg SBP or < 180 mmHg SBP. Treatment must be implemented as soon as possible after radiological confirmation of diagnosis. Antihypertensive therapy must begin within 6 hours of symptom onset. The patient will be re-imaged 24 hours later. The patient will have continuous non-invasive BP and heart rate(HR) monitoring for a minimum of 24 hours. Antihypertensive drug use and dosage will be recorded with BP and HR. Patients will be monitored regularly until study completion. MRI's will be done at 48 hours, day 7 and day 30. This imaging will help to detect ischemic changes that may occur. Blood will be collected at the same time as the MRI. Blood analysis will be done to possibly identify biomarkers that may be putative mediators of ischemic injury in ICH patients.

DETAILED DESCRIPTION:
Study Design: multi-centre randomized open-label, blinded-endpoint trial of two different BP management strategies. This study is being conducted in the Emergency Departments and Stroke Units of Canadian academic and non-academic centres.

Overall Aim and Hypothesis: The primary study aim is to assess the rate of ischemic lesion development in patients randomized to two different BP treatment strategies. The overall a priori hypothesis is that aggressive BP reduction will not be associated with ischemic injury after ICH.

Patients: Male and female patients will be recruited from Emergency Departments of participating hospitals. A total of 270 patients will be included over 3 years.

Baseline Data and Randomization: Demographics, Glasgow Coma Scale (GCS) and National Institutes of Health Stroke Scale (NIHSS) scores (both of which are part of routine stroke patient assessment), time of symptom onset and diagnostic CT scan will all be recorded. If the CT scan is completed within 6 hours of onset and confirms evidence of a primary ICH, patients will be randomized. Where patients are incompetent and surrogate decision makers are not immediately available, randomization will occur using a deferred consent procedure. Stroke risk factors, past medical history and medications, with emphasis on antihypertensives, as well as standard clinical blood work (complete blood count and coagulation profile) will be recorded after randomization in order to avoid delays to BP treatment.

Intervention - Blood Pressure Management Protocols:

"Aggressive" BP Target (<140 mmHg) Treatment Group: Patients randomized to the <140 mmHg group (n=135) will immediately receive a 10 mg IV bolus of labetalol, administered over 1 minute. A protocol designed to achieve and maintain systolic BP <140 mmHg within 60 minutes of randomization has been designed (Appendix 5). A key feature of this protocol is the utilization of IV enalapril, which can be given regularly (Q. 6 hourly), avoiding BP fluctuations, a problem which has been noted previously when using bolus-based protocols.109 Patients randomized to the <140 mmHg group will be treated with 1.25 mg of IV enalapril immediately after labetalol administration. A lower limit of 120 mmHg has been stipulated, although given the investigators experience in ICH ADAPT I, this is unlikely to be achieved. In the event of systolic BP falling below 120 mmHg, antihypertensive therapy will be held and patients will be fluid resuscitated with isotonic saline. Pressor agents will not be used.

"Conservative" BP Target (<180 mmHg) Treatment Group: Patients randomized to the <180 mmHg group (n=135) will be administered parenteral antihypertensive therapy only if systolic BP is ≥180 mmHg, consistent with current guidelines.

All patients will have continuous non-invasive BP and heart rate (HR) monitoring for a minimum of 24h. BP and HR will be recorded most intensively during the hyperacute phase, as per the NINDS r-tPA protocol for vital signs monitoring. Antihypertensive drug use and dosages will be recorded concomitantly with BP and HR. Patients will be monitored regularly until study completion. Door-to-needle times will be documented with respect to the initiation of antihypertensive medication and the proportion of patients achieving BP targets within 1 hour of treatment.

At completion of the 24h active treatment period, all patients will continue to receive standard stroke care and rehabilitation, and treating physicians will manage BP in the manner they feel is appropriate. Physicians will be encouraged to start oral antihypertensive therapy, administered via nasogastric feeding tube if necessary, on day 2. BP, HR and antihypertensive medication doses will continue to be monitored and recorded every 4 h for the first 48 h and then twice daily until discharge. Long-term goals for both patient groups after the active treatment period are a systolic BP of <140 mmHg, or <130 mmHg in those with diabetes, as per current stroke prevention and hypertension guidelines.

Imaging Procedures:

Baseline - Immediately prior to randomization and BP reduction, patients will undergo a standard non-contrast CT diagnostic brain scan. In the event of early neurological deterioration at any point, a repeat CT scan will be obtained immediately.

24 hour CT - All patients will have a repeat CT brain scan at 24±3 h, in order to assess for hematoma expansion and peri-hematoma edema volume.

48 hour MRI - At 48±12 h, patients will undergo MRI scanning, including a T1-weighted sagittal localizer, DWI, Gradient Recalled Echo (GRE)/Susceptibility Weighted Imaging (SWI), diffusion-weighted (DWI) and perfusion-weighted images (PWI).

Day 7 MRI Scan (Secondary Endpoint) - A repeat MRI will be obtained at 7±2 days to assess for new DWI lesion development and evolution of those identified at 24 hours.

Day 30 MRI Scan (Secondary Endpoint) - A repeat MRI will be obtained at 30±5 days to assess for new DWI lesion development and evolution of those identified at 24 hours and 7 days.

Clinical Assessments:

In Hospital - In addition to BP data, GCS and NIHSS scores will be collected in the event of early neurological deterioration. Both of these scores will also be recorded at the time of each MRI scan and at hospital discharge or transfer to alternate level of care, i.e. rehabilitation or long-term care facility. Discharge modified Rankin Scores (mRS) will also be recorded. Cognitive changes will be assessed with the Montreal Cognitive Assessment (MoCA) at the time of each MRI scan.

Follow-up (Day 30) - A standardized interview aimed at determining mortality and current residence of the patient (home/hospital/rehabilitation hospital/long-term care facility) will be administered at the time of the day 30 MRI. The NIHSS and MoCA scores will also be recorded, as will modified Rankin scale (mRS) scores. Quality of life will be assessed with the EQ-5D.

(Day 90) - This is the standard time point for measuring functional outcomes in stroke trials, as the bulk of neurological recovery occurs within that time frame. All neurological, functional and cognitive disability tests will be repeated at this time.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Acute primary ICH demonstrated with CT scan, within 6 h of symptom onset.
* Two systolic BP measurements ≥140 mmHg recorded >2 min apart to qualify for enrolment.
* Onset ≤ 24 h prior to randomization

Exclusion Criteria:

* Contraindication to BP reduction i.e., severe arterial stenosis or high-grade stenotic valvular heart disease
* Indication for urgent BP reduction i.e., hypertensive encephalopathy, or aortic dissection
* Definite evidence that the ICH is secondary to underlying cerebral or vascular pathology, i.e., AVM, aneurysm, tumour, trauma, vasculitis, or hemorrhagic transformation of an ischemic infarct
* Previous ischemic stroke within 90 days of current event NB: Prior ICH is not an exclusion criterion
* Patients with suspected secondary cause of ICH.
* Planned surgical resection of hematoma NB: Extraventricular Drain placement is not an exclusion criterion
* Contraindication to CT perfusion imaging (i.e. contrast allergy, metformin use or Creatinine >160 μmol/l)
* Patients with pre-existing disability and dependence (defined as a pre-morbid modified Rankin Scale score ≥3) will be excluded
* Patients with life expectancy <6 months due to pre-morbid conditions/terminal illness
* Patients with known definite contraindications to MRI (pacemaker, ferrous metallic foreign body)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2011-08-01 (Actual); Primary Completion 2021-11 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Diffusion-weighted imaging (DWI) lesion frequency | 48 hours

SECONDARY OUTCOMES:
Cumulative diffusion-weighted imaging (DWI) lesion frequency | 30 days post randomization
Absolute hematoma growth | 24 hours post randomization
Functional disability as assessed by the Modified Rankin Scale | 90 days post randomization
  Modified Rankin scale (0=no symptoms, 1=no significant disability, 2=slight disability, 3=moderate disability, 4=moderately severe disability, 5=severe disability, 6=dead)

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - Ottawa Hospital Research Institute, Ottawa, Ontario

REFERENCES:
- [Derived] Gioia L, Klahr A, Kate M, Buck B, Dowlatshahi D, Jeerakathil T, Emery D, Butcher K. The intracerebral hemorrhage acutely decreasing arterial pressure trial II (ICH ADAPT II) protocol. BMC Neurol. 2017 May 19;17(1):100. doi: 10.1186/s12883-017-0884-4. PMID 28525977